CLINICAL TRIAL: NCT07380724
Title: The Effect of Telehealth-Based Follow-Up on Functional Status, Self-Care Ability, and Activities of Daily Living in Patients Undergoing Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: The Effect of Tele-Health Application on Functional Status, Self-Care Ability and Activities of Daily Living in Individuals Undergoing Total Knee Arthroplasty Surgery
Acronym: (TKA-TELECARE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya Applied Sciences University (Other)
Responsible Party: Principal Investigator, Rümeysa Demir, Lecturer, Sakarya Applied Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SakaryaAppliedSciencesUni; 2024/4 (Other: University of Health Sciences)
Record Dates: First submitted 2025-07-30; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Arthroplasty; Telehealth; Self-Care Ability
Keywords: Functional Status, Activities of Daily Living, Self-Care Ability, Telehealth, Total Knee Arthroplasty
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Effect of Tele-Health Application on Functional Status, Self-Care Ability and Activities (Experimental): To investigate the effect of telehealth services on functional status, self-care ability, and activities of daily living after total knee arthroplasty.
  Interventions: Other: tele health

INTERVENTIONS:
Other: tele health — To investigate the effect of telehealth services on functional status, self-care ability, and activities of daily living after total knee arthroplasty.
  Other Names: telehealt

SUMMARY:
Osteoarthritis, defined as a degenerative joint disease, is a chronic, non-inflammatory condition characterized by deterioration of joint cartilage and new bone formation on joint surfaces and margins. Due to osteoarthritis, the number of total knee arthroplasty (TKA) procedures has increased. Patients undergoing TKA often experience difficulties in meeting their self-care needs and performing daily living activities due to impaired functional status. During the postoperative home care period, nursing support is critical in enhancing patients' functional status, self-care ability, and independence in daily activities. Therefore, this study aims to examine the effect of telehealth services on functional status, self-care ability, and daily living activities in patients undergoing TKA. The study is designed as a randomized controlled trial. The sample will consist of patients who undergo TKA in the Orthopedics and Traumatology Department of Sakarya University Training and Research Hospital between April 2024 and April 2025. Patients in the intervention group will receive telehealth-based nursing follow-up, including education and counseling for 14 days after discharge. The control group will receive only standard discharge education. Data will be collected using the Structured Patient Information Form, WOMAC Osteoarthritis Index, Self-Care Agency Scale, Barthel Index of Activities of Daily Living, Subcutaneous Heparin Injection Evaluation Form, and Telephone Interview Form. Based on power analysis, a total of 54 participants are needed to achieve 85% power at a 95% confidence level and medium effect size (p < 0.05). To account for potential data loss, the sample size was increased to 60. It is anticipated that utilizing telehealth services for postoperative nursing follow-up will contribute significantly to patient safety, healthcare costs, and the nursing discipline.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or older
* Undergoing primary total knee arthroplasty due to osteoarthritis
* Able to communicate verbally and use a telephone or mobile device
* Discharged to home (not transferred to rehabilitation or nursing facility)
* Volunteering to participate and providing informed consent
* Having cognitive competence to answer questionnaires and follow instructions
* Access to a mobile phone or internet connection at home for telehealth follow-up

Exclusion Criteria:

* Undergoing revision knee arthroplasty or bilateral knee arthroplasty
* Having significant hearing, visual, or cognitive impairment that interferes with communication
* Diagnosed with advanced neurological or psychiatric disorders
* Having a severe postoperative complication (e.g., deep infection, reoperation)
* Being enrolled in another intervention study simultaneously
* Residing in a long-term care facility or nursing home
* Unable or unwilling to participate in telehealth-based interventions

Ages: 40 Weeks to 90 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Change in functional status, as measured by the WOMAC Osteoarthritis Index, from baseline (pre-operative) to 14 days post-discharge. | From baseline (preoperative assessment) to 14 days after discharge
  Functional status will be assessed using the WOMAC Osteoarthritis Index, which evaluates pain, stiffness, and physical function. Scores will be recorded at baseline (before surgery) and at the end of a 14-day telehealth-based follow-up period post-discharge.

SECONDARY OUTCOMES:
Change in self-care ability measured by the Self-Care Agency Scale | From baseline (preoperative assessment) to 14 days after discharge
  Self-care ability will be assessed using the Self-Care Agency Scale. The scale evaluates the individual's capacity to meet their own self-care needs. Scores will be obtained before surgery and after the 14-day telehealth follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University of Applied Sciences, Sakarya, Akyazı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will not be shared because the study involves sensitive patient information and data confidentiality must be maintained in accordance with ethical and institutional guidelines.

REFERENCES:
- [Result] Tsang MP, Man GCW, Xin H, Chong YC, Ong MT, Yung PS. The effectiveness of telerehabilitation in patients after total knee replacement: A systematic review and meta-analysis of randomized controlled trials. J Telemed Telecare. 2024 Jun;30(5):795-808. doi: 10.1177/1357633X221097469. Epub 2022 May 12. PMID 35549756